CLINICAL TRIAL: NCT03514979
Title: Acquired Immunodeficiency in ANCA (Antineutrophil Cytoplasmic Antibody) Associated Vasculitis
Brief Title: Acquired Immunodeficiency in ANCA Associated Vasculitis
Acronym: ACQUIVAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Arthritis Research UK (Other)
Responsible Party: Principal Investigator, Dr. Rona Smith, Clinical lecturer in nephrology and experimental medicine, Cambridge University Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCTU0155
Record Dates: First submitted 2018-04-13; First posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Systemic Vasculitis
MeSH Terms: conditions — Systemic Vasculitis | interventions — 13-valent pneumococcal vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Intervention Model Description: This is a phase IIb, open label study to evaluate the responses of patients with ANCA associated vasculitis (AAV) to pneumococcal vaccination. It has been designed primarily to assess the immunogenicity of pneumococcal vaccines in patients with AAV treated with rituximab compared to disease controls, but also to provide mechanistic information on vaccine response by comparing AAV patients and healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AAV patients treated with rituximab (Experimental): Pneumococcal Polysaccharide Conjugate vaccination at Month 0 and then Pneumococcal Polysaccharide Vaccination at Month 6.
  Interventions: Biological: Pneumococcal Polysaccharide Conjugate vaccination and Pneumococcal Polysaccharide Vaccination
- AAV patients - never received rituximab (Experimental): Pneumococcal Polysaccharide Conjugate vaccination at Month 0 and then Pneumococcal Polysaccharide Vaccination at Month 6.
  Interventions: Biological: Pneumococcal Polysaccharide Conjugate vaccination and Pneumococcal Polysaccharide Vaccination
- Healthy controls (Experimental): Pneumococcal Polysaccharide Conjugate vaccination at Month 0 and then Pneumococcal Polysaccharide Vaccination at Month 6.
  Interventions: Biological: Pneumococcal Polysaccharide Conjugate vaccination and Pneumococcal Polysaccharide Vaccination

INTERVENTIONS:
Biological: Pneumococcal Polysaccharide Conjugate vaccination and Pneumococcal Polysaccharide Vaccination — Pneumococcal vaccines
  Other Names: Prevnar 13 and Pneumovax

SUMMARY:
This study will address the following hypothesis: Rituximab therapy leads to an acquired immune deficiency, as demonstrated by impaired vaccine responses, in AAV patients.

Aims:

1. To investigate whether rituximab leads to immune deficiency in patients with AAV when compared to both disease and healthy controls.
2. To investigate whether the degree of immune deficiency is associated with the degree of B cell depletion.
3. To investigate whether T-independent vaccine responses are more severely affected than T-dependent vaccine responses after rituximab and whether a conjugated vaccine will overcome this postulated deficit in T independent vaccine responses.

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial all participants must:

* Have given written informed consent to participate
* Be aged 40 years and over

For patients in Group 1 only (rituximab treated):

* Have a diagnosis of AAV [granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA) or eosinophilic granulomatosis with polyangiitis (eGPA)]
* Have current or historical PR3/MPO ANCA positivity by ELISA or histological confirmation of AAV
* Have received ≥ 2g rituximab
* Have received their last dose of rituximab at least 12 months prior to enrolment
* Be in stable remission with a prednisolone dose of ≤ 5mg/day

For patients in Group 2 only (disease controls who have never received rituximab):

* Have a diagnosis of AAV (GPA, MPA or eGPA)
* Have current or historical PR3/MPO ANCA positivity by ELISA or histological confirmation of AAV
* Have received cyclophosphamide (oral or IV) as initial induction therapy
* Be on stable immunosuppression for the 6 months preceding screening including prednisolone ≤ 5mg/day AND either azathioprine, methotrexate or mycophenolate mofetil (at stable or tapering dose)

For healthy controls:

• Healthy individuals aged 40 years and over

Exclusion Criteria:

The presence of any of the following will preclude participant inclusion:

* Age < 40 years
* History of severe allergic or anaphylactic reactions to pneumococcal vaccinations
* Pneumococcal vaccination within 5 years prior to screening
* Females who are pregnant, plan to become pregnant, or breast feeding
* Medical, psychiatric, cognitive or other conditions that, in the investigator's opinion, compromise the patient's ability to understand the patient information, give informed consent, comply with the trial protocol, or to complete the study.
* History of malignancy within the past five years or any evidence of persistent malignancy, except fully excised basal cell or squamous cell carcinomas of the skin, or cervical carcinoma in situ which has been treated or excised in a curative procedure.
* Replacement immunoglobulin (IVIg) administered intravenously or subcutaneously in the 12 weeks prior to screening visit.

For patients in Groups 1 and 2 only (AAV patients):

* Presence of another multisystem autoimmune rheumatic disease
* The prior receipt of more than 36g of cumulative cyclophosphamide ever (either IV or oral)

For patients in group 1 only (rituximab group)

• The receipt of any immune suppressing agent (azathioprine, methotrexate or mycophenolate mofetil) after rituximab

For patients in Group 2 only (disease controls):

* A relapse of AAV within the 6 months prior to screening which has necessitated an increase in prednisolone or azathioprine, methotrexate or MMF dose.
* Previous rituximab therapy at any time

For healthy controls:

* Any history of any autoimmune condition
* Any history of use of immune suppressing medication, including > 4 weeks of oral glucocorticoids, within the 5 years prior to screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportions of rituximab treated patients to disease controls who respond to the Pneumococcal Polysaccharide Conjugate vaccine. measured at 28 (+/- 7) days after administration of vaccine. | Measured at 28 (+/- 7) days after administration of vaccine.
  Response is defined as at least a twofold increase in immunoglobulins in at least 6/13 pneumococcal serotypes tested.

SECONDARY OUTCOMES:
Immunoglobulin (IgG) titres for each individual serotype in the pneumococcal vaccine | Measured at month 0, 1, 6 and 7 in all participants
  Immunoglobulin (IgG) titres for each individual serotype in the pneumococcal vaccine
Number of serious adverse events, and serious adverse events specifically related to the vaccines administered | 7 months: end of trial
  Number of serious adverse events, and serious adverse events specifically related to the vaccines administered
Incidence, type, severity and treatment of infections experienced by participants after vaccinations | 7 months: end of trial
  Incidence, type, severity and treatment of infections experienced by participants after vaccinations
Changes in immunoglobulin levels | 7 months: end of trial
  Changes in immunoglobulin levels